CLINICAL TRIAL: NCT03680612
Title: Randomized, Double-Blind, Multi-Center Study of Cefepime/AAI101 in Hospitalized Adults With Complicated Urinary Tract Infections, Including Acute Pyelonephritis
Brief Title: Cefepime/AAI101 Phase 2 Study in Hospitalized Adults With cUTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allecra (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-201
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cefepime; enmetazobactam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefepime 1G - 2G / AAI101 0.5G - 0.75G (Experimental): cefepime 1 g or cefepime 2 g in combination with AAI101 500 mg or 750 mg
  Interventions: Drug: Cefepime 1G - 2G / AAI101 0.5G - 0.75G
- cefepime monotherapy (Active Comparator): cefepime 1 g or cefepime 2 g
  Interventions: Drug: cefepime 1 g or cefepime 2 g

INTERVENTIONS:
Drug: Cefepime 1G - 2G / AAI101 0.5G - 0.75G — Experimental drug
  Other Names: cefepime/AAI101 combination
  Arms: Cefepime 1G - 2G / AAI101 0.5G - 0.75G
Drug: cefepime 1 g or cefepime 2 g — cefepime monotherapy
  Other Names: cefepime alone
  Arms: cefepime monotherapy

SUMMARY:
Phase 2, randomised, double-blind, 2-cohort study in hospitalised adults with complicated urinary tract infection (cUTI), including acute pyelonephritis. All study cohorts were randomised in a 2:1 ratio. Treatment duration for each cohort was 7 to 10 days. Patients were not permitted to switch to oral therapy.

Cohort 1: 15 patients treated with cefepime 1 g/AAI101 500 mg intravenous (i.v.) infusion over 2 hours once every 8 hours (q8h), and 7 patients treated with cefepime 1 g i.v. infusion over 2 hours q8h.

Cohort 2: 15 patients treated with cefepime 2 g/AAI101 750 mg i.v. infusion over 2 hours q8h, and 8 patients treated with cefepime 2 g i.v. infusion over 2 hours q8h.

ELIGIBILITY:
Inclusion criteria:

• Male or female patients with clinical signs and/or symptoms of cUTI or acute pyelonephritis that were expected to require hospitalization and initial treatment with at least 7 days of i.v.

antibiotics.

Exclusion criteria:

* Patients with concurrent infection that would interfere with evaluation of response to the study antibiotics;
* Patients needing concomitant systemic antimicrobial agents in addition to those designated in the various study treatment groups;
* Patients receiving effective antibacterial drug therapy for any indication for a continuous duration of >24 hours during the previous 72 hours before the study-qualifying baseline urine was obtained or receiving any amount of potentially therapeutic antibacterial therapy after collection of the pre-treatment baseline urine culture and before administration of the first dose of study drug;
* Patients likely to require the use of an antibiotic for cUTI or acute pyelonephritis prophylaxis during participation in the study;
* Patients with confirmed fungal urinary tract infection at the screening visit (with ≥103 fungal colony forming units [CFU]/mL); or
* Patients with intractable urinary infection at baseline that the Investigator anticipated would require >10 days of study drug therapy were excluded from participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Microbiological Response at the Test of Cure (TOC) Visit in the Microbiological Modified Intent-to-Treat (mMITT) Population | 6 to 9 days post-End of Treatment
  Microbiological response is eradication for each baseline pathogen

SECONDARY OUTCOMES:
Microbiological Response at the TOC Visit in the Microbiologically Evaluable (ME) Population. | 6 to 9 days post-End of Treatment
  Microbiological response is eradication for each baseline pathogen

CONTACTS AND LOCATIONS:
Locations (5):
- Kromerizska nemocnice, Kroměříž, Czechia
- Jahn Ferenc Del-pesti Korhaz, Budapest, Hungary
- Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Klinika Chorob Wewnetrznych, Nefrologii i Transplantologii, Warsaw, Poland
- Fakultna nemocnica s poliklinikou J.A. Reimana Presov, Prešov, Slovakia
- Chernihiv City Hospital #2 of Chernihiv City Council, department of Urology, Chernihiv, Ukraine

IPD SHARING:
Plan to Share IPD: No